CLINICAL TRIAL: NCT05815745
Title: Physiological vs Right Ventricular Pacing Outcome Trial Evaluated for bradyCardia Treatment
Brief Title: "Physiological vs Right Ventricular Pacing Outcome Trial Evaluated for bradyCardia Treatment" (PROTECT-HF)
Acronym: PROTECT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22HH7931
Record Dates: First submitted 2023-02-13; First posted 2023-04-18 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Bradycardia; Pacing; Right Ventricular Pacing; His Bundle Pacing; Left Bundle Branch Area Pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right ventricular pacing (Active Comparator): Right ventricular pacing (apical or septal lead locations as per the implanting physicians' normal practice)
  Interventions: Device: Pacemaker - Right Ventricular pacing
- Physiological pacing (Experimental): The approach for physiological pacing will be either His bundle pacing or left bundle pacing at the operator's discretion. If both of these are not achieved biventricular pacing will be performed.
  Interventions: Device: Pacemaker - Physiological pacing

INTERVENTIONS:
Device: Pacemaker - Physiological pacing — The approach for physiological pacing will be either His bundle pacing or left bundle pacing at the operator's discretion. If both of these are not achieved biventricular pacing will be performed.
  Arms: Physiological pacing
Device: Pacemaker - Right Ventricular pacing — Right ventricular pacing (apical or septal lead locations as per the implanting physicians' normal practice).
  Arms: Right ventricular pacing

SUMMARY:
The PROTECT-HF multi-centre randomised controlled trial will compare two different pacing approaches for treating patients with slow heart rates. In it the investigators will compare a long-standing standard approach for pacing; right ventricular pacing, with a new form of pacing, physiological pacing (His and Left bundle area pacing) in 2600 patients.

Patients will be allocated at random to receive either right ventricular pacing or physiological pacing. Endpoint measurements will be undertaken at baseline, and at six-monthly intervals post-randomisation. Treatment allocation will be blinded to the endpoint assessor and the patient.

Recruitment and pacemaker implantation will be carried out at each participating centre. The primary analysis will be intention to treat. The investigators will also perform an on-treatment analysis.

2048 patients are needed to detect the expected effect size with 85% power. A total of 2600 patients will be recruited to allow for patient drop-out and crossover.

500-patient sub-study will assess within patient, and between groups, echocardiographic changes over a 24-month period to try and improve mechanistic understanding of PICM (Pacing Induced Cardiomyopathy).

DETAILED DESCRIPTION:
Patients entering the study will attend for implantation of a pacemaker device and be randomised to either right ventricular pacing or physiological pacing.

Patients at sites participating in echo sub-study will be informed of and given opportunity to consent to echo sub-study, this will be optional to them, even if they have consented to the main study.

ELIGIBILITY:
We will recruit patients who are referred for clinically indicated pacemaker implantation

Inclusion Criteria:

1. Adults aged over 18 with left ventricular ejection fraction >35% and one or more of the following guideline based ventricular pacing indications:

1. Permanent or intermittent 3rd degree AV block
2. Permanent or intermittent Mobitz type II AV block
3. First Degree AV block with a pacing indication
4. Slow chronic Atrial Fibrillation or Proposed AV node ablation
5. Bifascicular block with a pacing indication
6. Trifascicular block with a pacing indication
7. Wenckebach with a pacing indication

Exclusion Criteria:

1. Patients who are likely to only need occasional ventricular pacing, i.e. those with isolated sick sinus syndrome.
2. Pregnant women.
3. Unable to provide informed consent.
4. Those with comorbidity leading to a life expectancy <1year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2600 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2029-12-04 (Estimated); Study Completion 2029-12-04 (Estimated)

PRIMARY OUTCOMES:
Mortality | From date of consent, until date of death from any cause, assessed up until 78 months.
  Death, any cause
Heart Failure Morbidity | From date of consent, assessed up until 78 months, or death from any cause, whichever came first.
  Adjudicated unplanned heart failure acute care (hospital admissions or ambulatory diuretic therapy i.e. diuretic lounge visit).

SECONDARY OUTCOMES:
Incidence of clinically indicated upgrade to conventional biventricular pacing (CRT device) | From date of randomisation until the date of first documented incident of device upgrade, or death from any cause, whichever came first, assessed up to 78 months.
Patient quality of life assessed via questionnaires (EQ-5D-5L) EQ-5D is the name of the instrument and is not an acronym. | From date of consent, assessed up to 78 months or until death of any cause, whichever came first.
  The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ 'visual analogue scale' (EQ VAS).
  The descriptive system is made up of 5 sections: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  A High score on the descriptive section means a worse health outcome. A Low score on the descriptive section means a better health outcome. A value set is required to convert the outcomes into scores.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative (numerical) measure of health outcome that reflect the patient's own judgement.
  A high score on the VAS means a better outcome. A low score on the VAS means a worse outcome.
Patient symptoms assessed on a scale of 0-100 monthly | From one month after device implant date, assessed up to 78 months or until death of any cause, whichever came first.
  This questionnaire will be sent to participants on a monthly basis for the duration of the study, 78 months from one month post pacemaker implant until end of study (78 months) or death from any cause, whichever came first.
Safety endpoints: Device infections (requiring device extraction), pacing thresholds, need for lead revision or reimplantation, generator change, haematoma and pneumothorax | From device implant date, assessed up to 78 months or until death of any cause, whichever came first.
Pacemaker derived endpoints: a) Atrial fibrillation (duration >6minutes) b) Ventricular arrhythmia incidence c) Daily patient activity (hours stratified by device vendor) | From device implant date, assessed up to 78 months or until death of any cause, whichever came first.
Patient quality of life assessed via questionnaires '36-Item Short Form Health Survey' (SF-36) | From date of consent, assessed up to 78 months or until death of any cause, whichever came first.
  A high score defines a more favourable health state. Range 0 to 100.
Echo Sub-Study Endpoint: Left Ventricular End Systolic Volume (LVESV) (>10mls) within group differences | From baseline echocardiogram (0 to 6 weeks post pacemaker implant) to follow-up echocardiogram (24±1 months post pacemaker implant).
  Within group differences of Left Ventricular End Systolic Volume (>10mls) for differences according to treatment allocation.
Echo Sub-Study Endpoint: Ejection Fraction (EF) within patient changes | From baseline echocardiogram (0 to 6 weeks post pacemaker implant) to follow-up echocardiogram (24±1 months post pacemaker implant).
  Within patient changes in Ejection Fraction will be assessed for differences according to treatment allocation.
Echo Sub-Study Endpoint: Left Ventricular End Systolic Volume (LVESV) (>10mls) within patient changes | From baseline echocardiogram (0 to 6 weeks post pacemaker implant) to follow-up echocardiogram (24±1 months post pacemaker implant).
  Within patient changes of Left Ventricular End Systolic Volume (>10mls) for differences according to treatment allocation
Echo Sub-Study Endpoint: Ejection Fraction (EF) within group differences | From baseline echocardiogram (0 to 6 weeks post pacemaker implant) to follow-up echocardiogram (24±1 months post pacemaker implant).
  Within group differences in Ejection Fraction will be assessed for differences according to treatment allocation.

CONTACTS AND LOCATIONS:
Locations (45):
- Beacon Hospital, Dublin, Ireland
- Univerisity Medical Centre Ljubljana, Ljubljana, Slovenia
- United Kingdom (43):
  - Aberdeen Royal Infirmary, Aberdeen
  - Queen's Hospital, Barking
  - Good Hope Hospital, Birmingham
  - Queen Elizabeth Hospital, Birmingham
  - University Hospital Dorset, Bournemouth
  - Royal SUSSEX County Hospital, Brighton
  - Bristol Heart Institute, Bristol
  - Royal Papworth Hospital, Cambridge
  - St Richard's Hospital, Chichester
  - University Hospital Coventry, Coventry
  - Croydon, Croydon
  - Royal Infirmary of Edinburgh, Edinburgh
  - Victoria Hospital, Fife Keith
  - Medway Maritime Hospital, Gillingham
  - Wycombe Hospital, High Wycombe
  - Forth Valley Royal Hospital, Larbert
  - Leeds Teaching Hospital, Leeds
  - Glenfield Hospital, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Hammersmith Hospital, London
  - Kettering Hospital, London
  - King's College Hospital, London
  - Royal Free London/ Barnet Hospital, London
  - St Bartholomew's Hospital, London
  - Watford General Hospital, London
  - James Cook Hospital, Middlesbrough
  - King's Mill Hospital, Nottingham
  - Nottingham City Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Queen Alexandra Hospital, Portsmouth
  - Royal Berkshire, Reading
  - East Surrey, Redhill
  - Rotherham General Hospital, Rotherham
  - Northern General, Sheffield
  - Wexham Park Hospital, Slough
  - Southampton, Southampton
  - Morriston Hospital, Swansea
  - Great Western, Swindon
  - Musgrove Park Hospital, Taunton
  - Torbay Hospital, Torquay
  - UHS Worthing, Worthing
  - York Hospital, York

DOCUMENTS (1):
  • Study Protocol: Protocol_v9.0_16.06.2025 (2025-06-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT05815745/Prot_004.pdf